CLINICAL TRIAL: NCT01842607
Title: A Multi-centre, Open-label, Long-term Safety Study of Mepolizumab in Asthmatic Subjects Who Participated in theMEA115588 or MEA115575 Trials
Brief Title: A Study to Determine Long-term Safety of Mepolizumab in Asthmatic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115661
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: eosinophils; mepolizumab; SB-240563; safety; extension study; Severe refractory asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mepolizumab Arm (Experimental): Subjects will receive 100 mg of Mepolizumab (in polypropylene syringe) injected subcutaneously (SC) once every 4 weeks for 12 months
  Interventions: Biological: Mepolizumab

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab (a fully humanised IgG antibody) 100 mg injected SC once every 4 weeks for 12 months. Mepolizumab will be provided as a lyophilised cake in sterile vials

SUMMARY:
This is a multi-centre, open-label long-term safety study of 100 milligram (mg) mepolizumab administered subcutaneously (SC) every 4 weeks for 12 months in addition to standard of care in subjects who have severe, refractory asthma and a history of eosinophilic inflammation. Subjects who completed either MEA115588 or MEA115575 will be offered the opportunity to consent for this study.

ELIGIBILITY:
Inclusion Criteria:

* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Informed Consent: Prior to commencing any study related activities, subjects must be able and willing to provide written informed consent.
* MEA115588 or MEA115575 study completion: Completion of the double-blind investigational product treatment during MEA115588 or MEA115575.
* Current Anti-Asthma Therapy: Asthma is currently being treated with a controller medication (i.e., inhaled corticosteroids [ICS] or other asthma controlled medication) and the subject has been on a controller medication for the past 12 weeks. Subjects will be expected to continue controller therapy for the duration of the study.
* Male or eligible female subjects:
* To be eligible for entry into the study, females of childbearing potential must commit to consistent and correct use of an acceptable method of birth control for the duration of the trial and for 4 months after the last study drug administration.
* A serum pregnancy test is required of all females at the initial Baseline Visit (Visit 1). In addition, a urine pregnancy test will be performed for all females prior to enrollment, during each scheduled study visit prior to the injection of investigational product, and during the Follow-up Visit.

Exclusion Criteria:

* Hypersensitivity: Hypersensitivity reaction related to study medication during the MEA115588 or MEA115575 that led to patient withdrawal. Subjects who experienced a localized injection site reaction do not need to be excluded.
* Health Status: Clinically significant change in health status during MEA115588 or MEA115575 which in the opinion of the investigator would make the subject unsuitable for participation in this long-term study.
* Malignancy: A current malignancy or malignancy that developed during MEA115588 or MEA115575 (subjects that had localized carcinoma of the skin which was resected for cure will not be excluded). [Note for South Korea: Korean subjects with a diagnosis of malignancy within 5 years are excluded]
* Prior SAE: A study related SAE in MEA115588 or MEA115575 that was assessed as possibly related to study medication by the investigator.
* Pregnancy: Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* ECG: Baseline ECG which has a clinically significant abnormality or which shows corrected QT interval with Fridericia (QTcF) >=450 millisecond (msec) or QTcF >=480 msec for subjects with Bundle Branch Block.
* Smoking status: Current smokers
* Liver Function: Liver function tests that meet any of the following during one of the last treatment visits in MEA115588 or MEA115575 : alanine transaminase (ALT) >=2 x upper limit of normal (ULN); aspartate transaminase (AST) >=2 x ULN; alkaline phosphatase >=2 x ULN; Bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%
* Hepatitis Status: Positive Hepatitis B Surface Antigen (HBsAg) screen at Visit 1
* ECG Over-read: Clinically significant abnormality identified during the central over-read during one of the last treatment visits in MEA115588 or MEA115575

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2013-05-27 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (120):
- United States (19):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (4):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (3):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- France (10):
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Strasbourg
- Germany (11):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (8):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Pietra Ligure (SV), Liguria
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Cittadella (PD), Veneto
- Japan (12):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leeuwarden
- Poland (2):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
- Russia (3):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (9):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Donggu Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (3):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
- Ukraine (4):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (7):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Gibson PG, Prazma CM, Chupp GL, Bradford ES, Forshag M, Mallett SA, Yancey SW, Smith SG, Bel EH. Mepolizumab improves clinical outcomes in patients with severe asthma and comorbid conditions. Respir Res. 2021 Jun 7;22(1):171. doi: 10.1186/s12931-021-01746-4. PMID 34098955
- [Derived] Yancey SW, Ortega HG, Keene ON, Bradford ES. Efficacy of add-on mepolizumab in adolescents with severe eosinophilic asthma. Allergy Asthma Clin Immunol. 2019 Sep 3;15:53. doi: 10.1186/s13223-019-0366-x. eCollection 2019. PMID 31507641
- [Derived] Khurana S, Brusselle GG, Bel EH, FitzGerald JM, Masoli M, Korn S, Kato M, Albers FC, Bradford ES, Gilson MJ, Price RG, Humbert M. Long-term Safety and Clinical Benefit of Mepolizumab in Patients With the Most Severe Eosinophilic Asthma: The COSMEX Study. Clin Ther. 2019 Oct;41(10):2041-2056.e5. doi: 10.1016/j.clinthera.2019.07.007. Epub 2019 Aug 22. PMID 31447130
- [Derived] Ortega HG, Meyer E, Brusselle G, Asano K, Prazma CM, Albers FC, Mallett SA, Yancey SW, Gleich GJ. Update on immunogenicity in severe asthma: Experience with mepolizumab. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2469-2475.e1. doi: 10.1016/j.jaip.2019.03.042. Epub 2019 Apr 5. No abstract available. PMID 30954640
- [Derived] Lugogo N, Domingo C, Chanez P, Leigh R, Gilson MJ, Price RG, Yancey SW, Ortega HG. Long-term Efficacy and Safety of Mepolizumab in Patients With Severe Eosinophilic Asthma: A Multi-center, Open-label, Phase IIIb Study. Clin Ther. 2016 Sep;38(9):2058-2070.e1. doi: 10.1016/j.clinthera.2016.07.010. Epub 2016 Aug 21. PMID 27553751
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an extension of MEA115588 (NCT01691521) and MEA115575 (NCT01691508). Participants who completed the prior studies were offered to enroll in this study. Assessments that were captured as part of exit visit for MEA115588 and MEA115575 served as Baseline visit for this study.
Pre-assignment Details: 651 participants who completed the study MEA115588 or MEA115575 were enrolled in this study. Participants meeting all the inclusion criteria and none of the exclusion criteria received their first mepolizumab dose at Visit 1 and continued to receive mepolizumab subcutaneous (SC) injections approximately every 4 weeks for 12 months.
Groups:
- Mepolizumab 100 mg SC: Participants received mepolizumab 100 milligrams (mg) administered via subcutaneous (SC) injection into the upper arm or thigh approximately every 4 weeks for 12 months. Participants remained on standard of care asthma therapy which could be adjusted during the study at the discretion of the physician.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg SC
Started | 651
Completed | 585
Not Completed | 66
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 19
Not completed — Protocol Violation | 8
Not completed — Protocol defined stopping criteria | 2
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 9
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360
  Male | 291
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 14
  American Indian or Alaskan Native | 2
  Asian - Central/South Asian Heritage | 3
  Asian - East Asian Heritage | 44
  Asian - Japanese Heritage | 45
  Asian - South East Asian Heritage | 7
  Native Hawaiian or Other Pacific Islander | 1
  White - Arabic/North African Heritage | 13
  White - White/Caucasian/European Heritage | 517
  Mixed Race | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Including Both Systemic (i.e. Allergic/Immunoglobulin (Ig)E-mediated and Non-allergic) and Local Site Reactions
Description: AEs were collected from the Baseline visit until the follow-up visit (approx. 12 weeks post-last dose). Participants were monitored to evaluate the AEs of systemic and local site reaction. AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. On treatment AEs were defined as events occurring from the first dose until 28 days after the last dose of mepolizumab.
Time Frame: From Baseline visit until the follow-up visit (approximately [approx.] week 60 [12 weeks post-last dose])
Population: As Treated (AT) Population: all participants who received at least one dose of open label mepolizumab.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Any AEs | 558
  AEs related to study treatment | 119
  Any SAEs | 94
  SAEs related to study treatment | 1
  Fatal SAEs | 0

2. Secondary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies and Neutralizing Antibodies (NAb) at the Indicated Time Points
Description: Blood samples were collected for the determination of anti-mepolizumab antibodies (ADA) just prior to administration of mepolizumab at indicated time points. Samples that tested positive for anti-mepolizumab antibodies were further tested for the presence of NAb. Participants who switched from the 250 mg vial to the 100 mg vial required one immunogenicity sample prior to the first dose from the 100 mg vial and one sample prior to the second dose from the 100 mg vial at the next visit. The highest value post-baseline visit are based on each participant's highest post-baseline titer. NAb assay result was only presented for participants with positive ADA assay. Highest value post-baseline would be positive for a participant who had both negative and positive post-baseline results.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population. Only those participants available at the indicated timepoints were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Highest value post-baseline, ADA, positive, n=646 | 31
  Highest value post-baseline, ADA, negative, n=646 | 615
  Highest value post-baseline, NAb, positive, n=31 | 0
  Highest value post-baseline, NAb, negative, n=31 | 31

3. Secondary Outcome: Annualized Rate of Exacerbations Per Year
Description: Exacerbations are defined as the worsening of asthma which requires use of systemic corticosteroids (IV or oral steroid like prednisone, for at least 3 days or a single intramuscular (IM) corticosteroid (CS) dose is required. For maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visit. Analysis of the number of exacerbations was performed using a negative binomial model with covariates of region, exacerbations in the year prior to the start of MEA115588 or MEA115575 (as an ordinal variable) and baseline percent (%) predicted forced expiratory volume in 1 second (FEV1), and with logarithm of time on treatment as an offset variable.
Time Frame: Baseline up to Exit Visit (approx. 52 weeks) or if Early Withdrawal 4 weeks post last dose
Population: AT Population
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Exacerbations per year | 0.93 [0.83 to 1.04]

4. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire (ACQ) Score
Description: The ACQ-5 is a five-item questionnaire developed as a measure of participants asthma control. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, shortness of breath, wheeze). The response options for all these questions consist of a 0 (no impairment/limitation) to 6 (total impairment/ limitation) scale. The overall ACQ score is calculated as the mean of the 5 questions and therefore ranges between 0 (totally controlled) and 6 (severely uncontrolled). The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population, Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Score on scale
  Week 4, n=603 | -0.09 (0.812)
  Week 16, n=592 | -0.11 (0.920)
  Week 28, n=577 | -0.05 (1.021)
  Week 40, n=564 | -0.10 (0.944)
  Week 52, n=556 | -0.09 (0.990)
  Follow-up visit, n=338 | 0.20 (1.132)

5. Secondary Outcome: Mean Change From Baseline in Clinic Pre-bronchodilator FEV1 Over the 52-week Treatment Period
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry at Baseline, Week 16, Week 28 and Week 52. Spirometry was performed within ± 1 hour of the Baseline assessment. The change from Baseline is defined as the difference between the value of the end point at the time point of interest and Baseline value.
Time Frame: From Baseline and up to Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Milliliters (mL)
  Week 16, n=632 | 67 (362.7)
  Week 28, n=615 | 50 (409.8)
  Week 52, n=602 | 29 (406.2)

6. Secondary Outcome: Number of Participants Withdrawn Due to Lack of Efficacy and Adverse Events From the Study
Description: AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Withdrawals due to lack of efficacy | 19
  Withdrawals due to adverse events | 11

7. Secondary Outcome: Number of Participants Hospitalized Due to Exacerbations and Adverse Events
Description: AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Exacerbation is defined as worsening of asthma which requires use of systemic corticosteroids (IV or oral steroid like prednisone, for at least 3 days or a single intramuscular (IM) corticosteroid (CS) dose is required. For maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visit.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  No hospitalisation due to exacerbations | 612
  One time hospitalisation due to exacerbations | 29
  Two times hospitalisation due to exacerbations | 4
  Three times hospitalisation due to exacerbations | 4
  Four times hospitalisation due to exacerbations | 0
  Five times hospitalisation due to exacerbations | 0
  Six times hospitalisation due to exacerbations | 1
  Seven times hospitalisation due to exacerbations | 0
  Eight times hospitalisation due to exacerbations | 0
  Nine times hospitalisation due to exacerbations | 0
  Ten times hospitalisation due to exacerbations | 1
  No hospitalisation due to AEs | 560
  One time hospitalisation due to AEs | 61
  Two times hospitalisation due to AEs | 13
  Three times hospitalisation due to AEs | 11
  Four times hospitalisation due to AEs | 4
  Five times hospitalisation due to AEs | 0
  Six times hospitalisation due to AEs | 1
  Seven times hospitalisation due to AEs | 0
  Eight times hospitalisation due to AEs | 0
  Nine times hospitalisation due to AEs | 0
  Ten times hospitalisation due to AEs | 0
  Eleven times hospitalisation due to AEs | 0
  Twelve times hospitalisation due to AEs | 0
  Thirteen times hospitalisation due to AEs | 0
  Fourteen times hospitalisation due to AEs | 0
  Fifteen times hospitalisation due to AEs | 0
  Sixteen times hospitalisation due to AEs | 1

8. Secondary Outcome: Number of Participants With Systemic (i.e., Allergic/IgE-mediated and Non-allergic) and Local Site Reactions
Description: Participants were monitored to evaluate the AEs of systemic and local site reaction. AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Hypersensitivity reactions (i.e., allergic or IgE-mediated reactions) were monitored using the diagnostic criteria for anaphylaxis as outlined by the 2006 Joint NIAID/FAAN Second Symposium on Anaphylaxis. Information was also collected to assess localized site reactions as determined by the investigator. On treatment AEs were defined as events occurring from the first dose until 28 days after the last dose of mepolizumab.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Any systemic infusion/injection site reaction | 13
  Injection related reaction | 7
  Hypersensitvity | 4
  Type IV hypersensitivity reaction | 3
  Any local infusion/injection site reaction | 29

9. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings at Any Time Post Baseline
Description: 12-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. The ECG was obtained before lung function testing followed by other study procedures. ECG was performed at Baseline, Week 28, Week 52 and at the end of follow-up period (approx. 12 weeks post-last dose). ECG findings were summarised at any time post Baseline for participants as normal, abnormal-not clinically significant(A-NCS) and abnormal-clinically significant (A-CS).
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population, only participants with ECG results post-baseline were analyzed
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 638
Participants
  Normal | 262
  A-NCS | 295
  A-CS | 81

10. Secondary Outcome: Mean Change From Baseline in QT Interval Corrected by Bazett's Method (QTcB) and QT Interval Corrected by Fridericia's Method (QTcF) Values for ECG Assessed at Baseline, Week 28, Week 52 and at Follow-up Visit (Approx. 12 Weeks Post-last Dose)
Description: 12-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. The ECG was obtained before lung function testing followed by other study procedures. ECG was performed at Baseline, Week 28, Week 52 and at the end of follow-up period (approx. 12 weeks post-last dose). The change from Baseline is defined as the difference between the value of the end point at the time point of interest and Baseline value.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Milliseconds (msec)
  QTcB, Week 28, n=592 | -5.5 (19.10)
  QTcB, Week 52, n=573 | -3.2 (18.90)
  QTcB, Follow-up, n=299 | -3.4 (19.67)
  QTcF, Week 28, n=592 | -7.1 (16.15)
  QTcF, Week 52, n=573 | -3.5 (15.68)
  QTcF, Follow-up, n=299 | -5.5 (17.01)

11. Secondary Outcome: Number of Participants With Maximum Change From Baseline in QTcF Interval for ECG Assessed at Any Time Post Baseline
Description: 12-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. ECG was performed at Baseline, Week 28, Week 52 and at the end of follow-up period (approx. 12 weeks post-last dose). Participants with maximum change (MC) from Baseline were summarised at any time post Baseline for the following categories <-60, >=-60 to <-30, >=-30 to <0, >=0 to <30, >=30 to <60 and >=60. The change from Baseline is defined as the difference between the value of the end point at the time point of interest and Baseline value. QTc intervals shown at any time post Baseline are the maximum seen in each participant over the course of the trial.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 614
Participants
  MC <-60, n=614 | 2
  MC >=-60 to <-30, n=614 | 11
  MC >=-30 to <0, n=614 | 252
  MC >=0 to <30, n=614 | 328
  MC >=30 to <60, n=614 | 20
  MC >=60, n=614 | 1

12. Secondary Outcome: Number of Participants With Maximum Change From Baseline in QTcB Interval for ECG Assessed at Any Time Post Baseline
Description: 12-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. ECG was performed at Baseline, Week 28, Week 52 and at the end of follow-up period (approx. 12 weeks post-last dose). Participants with maximum change (MC) from Baseline were summarized at any time post Baseline for the following categories <-60, >=-60 to <-30, >=-30 to <0, >=0 to <30, >=30 to <60 and >=60. The change from Baseline is defined as the difference between the value of the end point at the time point of interest and Baseline value. QTc intervals shown at any time post Baseline are the maximum seen in each participant over the course of the trial. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 614
participants
  MC <-60, n=614 | 3
  MC >=-60 to <-30, n=614 | 16
  MC >=-30 to <0, n=614 | 222
  MC >=0 to <30, n=614 | 330
  MC >=30 to <60, n=614 | 41
  MC >=60, n=614 | 2

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure Assessed at Week 52
Description: Vital sign measurements including systolic blood pressure (SBP) and diastolic blood pressure (DBP) were performed at Baseline, at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and follow-up visit (approx. 12 weeks post-last dose). Vital measurements were done pre-injection with the participants sitting, having rested in this position for at least 5 minutes before each reading. They were taken before measurement of any clinic lung function tests or ECGs at the specified time point.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 581
Millimeter of mercury (mmHg)
  SBP, Week 52, n=581 | 0.3 (12.90)
  DBP, Week 52, n=581 | -0.4 (9.47)

14. Secondary Outcome: Change From Baseline in Pulse Rate Assessed at Week 52
Description: Vital sign measurements including sitting pulse was performed at Baseline, at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and follow-up visit (approx. 12 weeks post-last dose). Vital measurements were done pre-injection with the participants sitting, having rested in this position for at least 5 minutes before each reading. They were taken before measurement of any clinic lung function tests or ECGs at the specified time point.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Beats per minute (BPM) | 0.2 (10.52)

15. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters Outside the Normal Range at Any Time Post-baseline
Description: Clinical chemistry laboratory parameters included alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, calcium, chloride, cholesterol, creatine kinase, creatinine, direct bilirubin, gamma glutamyl transferase, high density lipoprotein (HDL) cholesterol, indirect bilirubin, low density lipoprotein (LDL) cholesterol, lactate dehydrogenase, phosphate, plasma/serum protein, potassium, serum glucose, sodium, triglycerides, urea, and very low density lipoprotein (VLDL) cholesterol assessed at the indicated time points. Laboratory abnormalities outside the normal range (high and low values) at any time post baseline were presented. Any time post Baseline = all visits (including scheduled and unscheduled). If participant had given both high and low value at least once then participant is counted under both high and low category for this visit.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: AT Population, Only those participants available at the specified time points were analyzed ( n=X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Alanine aminotransferase, High, n=649 | 70
  Albumin, Low, n=649 | 1
  Albumin, High, n=649 | 23
  Alkaline phosphatase, High, n=649 | 37
  Aspartate aminotransferase, High, n=649 | 53
  Bilirubin, High, n=649 | 38
  Calcium, Low, n=649 | 19
  Calcium, High, n=649 | 49
  Chloride, Low, n=649 | 9
  Chloride, High, n=649 | 126
  Cholesterol, High, n=649 | 492
  Creatine kinase, High, n=649 | 178
  Creatinine, Low, n=649 | 170
  Creatinine, High, n=649 | 18
  Direct bilirubin, High, n=649 | 10
  Gamma glutamyl transferase, High, n=649 | 146
  HDL cholesterol, Low, n=616 | 22
  Indirect bilirubin, High, n=649 | 12
  LDL cholesterol, High, n=604 | 207
  Lactate dehydrogenase, High, n=649 | 36
  Phosphate, Low, n=649 | 149
  Phosphate, High, n=649 | 84
  Plasma/serum protein, Low, n=649 | 29
  Potassium, Low, n=649 | 24
  Potassium, High, n=649 | 22
  Serum glucose, Low, n=649 | 62
  Serum glucose, High, n=649 | 239
  Sodium, Low, n=649 | 25
  Sodium, High, n=649 | 9
  Triglycerides, High, n=617 | 102
  Urea, Low, n=649 | 17
  Urea, High, n=649 | 53
  VLDL cholesterol, Low, n=605 | 13
  VLDL cholesterol, High, n=605 | 99

16. Secondary Outcome: Number of Participants With Haematology Laboratory Parameters Outside the Normal Range at Any Time Post-baseline
Description: Haematology laboratory parameters included basophils, basophils/leukocytes, blood erythrocytes, blood leukocytes, eosinophils, eosinophils/leukocytes, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), erythrocytes distribution width (EDW), hematocrit, hemoglobin, lymphocytes, lymphocytes/leukocytes, monocytes, monocytes/leukocytes, neutrophils segmented (NS), neutrophils/leukocytes, platelets, reticulocytes assessed at Baseline, Week 4, Week 16, Week 28, Week 52 and follow-up visit (approx. 12 weeks post-last dose). Hematology abnormalities outside the normal range (high and low values) at any time post baseline were presented. Any time post Baseline is equal to all visits (including scheduled and unscheduled) post Baseline were considered for this visit derivation. If participant had given both high and low value at least once then participant is counted under both high and low category for this visit.
Time Frame: From Baseline visit until the follow-up visit (approx. week 60 [12 weeks post-last dose])
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 651
Participants
  Basophils, High, n=649 | 2
  Basophils/Leukocytes, High, n=649 | 3
  Blood Erythrocytes, Low, n=649 | 52
  Blood Erythrocytes, High, n=649 | 36
  Blood Leukocytes, Low, n=649 | 25
  Blood Leukocytes, High, n=649 | 146
  Eosinophils, Low, n=649 | 429
  Eosinophils, High, n=649 | 51
  Eosinophils/Leukocytes, High, n=649 | 60
  MCHC, Low, n=649 | 276
  MCH, Low, n=649 | 58
  MCH, High, n=649 | 26
  MCV, Low, n=649 | 32
  MCV, High, n=649 | 32
  EDW, High, n=649 | 322
  Hematocrit, Low, n=649 | 57
  Hematocrit, High, n=649 | 94
  Hemoglobin, Low, n=649 | 116
  Hemoglobin, High, n=649 | 14
  Lymphocytes, Low, n=649 | 48
  Lymphocytes, High, n=649 | 25
  Lymphocytes/Leukocytes, Low, n=649 | 168
  Lymphocytes/Leukocytes, High, n=649 | 68
  Monocytes, Low, n=649 | 156
  Monocytes, High, n=649 | 15
  Monocytes/Leukocytes, High, n=649 | 45
  NS, Low, n=649 | 31
  NS, High, n=649 | 151
  Neutrophils/Leukocytes, Low, n=649 | 39
  Neutrophils/Leukocytes, High, n=649 | 226
  Platelets, Low, n=649 | 8
  Platelets, High, n=649 | 58
  Reticulocytes, Low, n=649 | 77
  Reticulocytes, High, n=649 | 294

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were collected from the first dose of study treatment until 28 days after the last dose of mepolizumab up to 52 weeks.
Description: Serious adverse events (SAEs) and Non-serious AEs were collected in members of As-Treated (AT) Population, comprised of all participants who received at least one dose of open label mepolizumab medication.
Arm/Group | Mepolizumab 100 mg SC
Serious Adverse Events (participants affected / at risk) | 94/651
Other Adverse Events (participants affected / at risk) | 461/651
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100 mg SC (N=651)
Asthma (Respiratory, thoracic and mediastinal disorders) | 38
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 4
Appendicitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Aspergillus infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Pharyngeal abscess (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyskinesia oesophageal (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Atrial fibrillation (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Type IV hypersensitivity reaction (Immune system disorders) | 1
Depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Nephrocalcinosis (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Retinal detachment (Eye disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Ejection fraction decreased (Investigations) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100 mg SC (N=651)
Nasopharyngitis (Infections and infestations) | 196
Upper respiratory tract infection (Infections and infestations) | 99
Bronchitis (Infections and infestations) | 78
Sinusitis (Infections and infestations) | 66
Influenza (Infections and infestations) | 28
Lower respiratory tract infection (Infections and infestations) | 26
Rhinitis (Infections and infestations) | 23
Urinary tract infection (Infections and infestations) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 46
Arthralgia (Musculoskeletal and connective tissue disorders) | 44
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21
Asthma (Respiratory, thoracic and mediastinal disorders) | 61
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Headache (Nervous system disorders) | 87
Injection site reaction (General disorders) | 29
Fatigue (General disorders) | 24
Nausea (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.